CLINICAL TRIAL: NCT06922162
Title: Behavioural and Physiological Responses to Tickling in Patients With Disorders of Consciousness
Brief Title: Tickle Stimulation in Disorders of Consciousness (DoC)
Acronym: TICKLING-DOC
Status: Recruiting | Type: Observational
Sponsor: Anna Estraneo (Other)
Responsible Party: Sponsor-Investigator, Anna Estraneo, MD Neurologist Senior researcher, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Other Study IDs: TICKLING-DOC
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Disorders of Consciousness
Keywords: Tickle stimulation; Behavioural evaluation; Neurophysiological evaluation; Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Neurophysiological Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with Disorders of Consciousness (DoC): All patients with disorders of consciousness who are consecutively admitted to the participating centers of the study will be enrolled with a diagnosis of disorders of consciousness based on the CRS-R scale, with an age ≥18 years and a time since the event ≥ 28 days.
  Interventions: Behavioral: Tickle stimulation; Device: Neurophysiological Monitoring with SedLine

INTERVENTIONS:
Behavioral: Tickle stimulation — Patients will be subjected to tickling:
  they will be tickled bilaterally in three areas, the soles of the feet, the armpits, and the ribs-plus a control area, the forehead. The stimulation will be manual and performed by rubbing the targeted body part while opening and closing the fingers in pairs in an arched motion. Additionally, patients will also undergo a neutral stimulation (in the same body areas), which consists of simply touching the area without inducing tickling.
Device: Neurophysiological Monitoring with SedLine — SedLine is a portable, non-invasive EEG monitoring device used to record electrical brain activity through frontal electrodes. In the TICKLING-DOC study, SedLine is used to assess cortical responses in patients with disorders of consciousness (DoC) during manual tactile stimulation, specifically tickling, and neutral touch. The EEG data are recorded before, during, and after stimulation to detect neural reactivity and possible correlations with behavioral responses. The goal is to investigate whether tickle-evoked EEG activity reflects residual consciousness and contributes to diagnostic and rehabilitative strategies. SedLine allows continuous monitoring in a bedside setting, offering safe, real-time assessment of brain function.
  Other Names: SedLine EEG Monitor; Masimo SedLine

SUMMARY:
The aim of this project is to investigate whether tickling stimulations can have a short-term effect on the responsiveness of patients with Disorders of Consciousness due to Severe Acquired Brain Injury and to compare this effect with that of neutral tactile stimulations that do not induce tickling.

DETAILED DESCRIPTION:
During the experimental session, patients will undergo the CRS-R and the Nociception Coma Scale-Revised (NCS-R) to ensure that any responses to tickling are not influenced by pain sensations. Subsequently, fNIRS detection optodes will be placed using a non-invasive frontal headband. A 10-minute resting-state recording will be performed. Next, patients will be subjected to tickling: they will be tickled bilaterally in the three most ticklish areas identified in a pilot study with healthy subjects-namely, the soles of the feet, the armpits, and the ribs-plus a control area, the forehead. The stimulation will be manual and will be performed by rubbing the targeted body part while opening and closing fingers in pairs in an arched motion. Additionally, patients will also receive a neutral stimulation (in the same body areas), which consists of simply touching the area without inducing tickling. The order of stimulations will follow a randomized list. Each stimulation will last for 5 seconds, followed by 5 seconds of rest, repeated twice. In total, patients will be stimulated for 10 seconds plus 5 seconds of rest (15 seconds in total) for each body area. There will be a 1-minute pause between each area. Afterward, an additional 10 minute resting-state fNIRS recording will be conducted. During the experimental session, patients will be filmed so that the videos can be analyzed by two different experimenters, who will assess differences between stimulations based on facial expressions, verbalizations/vocalizations, body movements, and changes in emotional state (e.g., crying, smiling, grimacing). At the end of the protocol, the fNIRS optodes will be removed. In total, the experiment will last approximately one hour and fifteen minutes: 30 minutes for CRS-R/NCS-R and 45 minutes for the tickling protocol and fNIRS recording.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of disorders of consciousness (DoC) based on the CRS-R scale;
* Age ≥18 years;
* Time since the event ≥ 28 days

Exclusion Criteria:

* Large craniectomy that may interfere with fNIRS recording; Unstable clinical conditions (e.g., respiratory failure, fever, status epilepticus, etc.);
* Fractures, paralysis, injuries, or muscular dystrophy that prevent proper stimulation of the aforementioned body parts;
* Lack of informed consent from the legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with DoC who are consecutively admitted to the participating centers of the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral Response Scores During Tickling and Neutral Stimulation (Video Coding) | Day 1 (single session)
  Behavioral responses will be evaluated from video recordings by two blinded raters, based on predefined observational categories (e.g., facial expressions, vocalizations, etc).
Hemodynamic Response Changes Measured by fNIRS During Tickling and Neutral Stimulation | Day 1 (single session)
  Oxygenated and deoxygenated hemoglobin changes (HbO/HbR) will be recorded using functional near-infrared spectroscopy (fNIRS) in response to tactile stimulation. Signal changes in prefrontal regions will be analyzed and compared across stimulation types.
Cortical EEG Activation Patterns During Tickling and Neutral Stimulation (SedLine) | Day 1 (single session)
  EEG data will be acquired with SedLine during stimulation sessions. Spectral power in defined frequency bands (e.g., alpha, beta) will be analyzed and compared between conditions.

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) Total Score Prior to Tickling Stimulation | Day 1 (baseline)
  Coma Recovery Scale-Revised (CRS-R) total score assessed before the stimulation protocol to determine baseline level of consciousness.The Coma Recovery Scale-Revised (CRS-R) is a standardized behavioral assessment tool used to determine the level of consciousness in patients with disorders of consciousness.
  Scores range from 0 to 23, with higher scores indicating better consciousness and functional responsiveness.
Nociception Coma Scale-Revised (NCS-R) Total Score Prior to Stimulation | Day 1 (baseline)
  NCS-R will be administered before tactile stimulations to assess nociceptive reactivity. The Nociception Coma Scale-Revised (NCS-R) is a standardised behavioural tool used to assess nociceptive responses in patients with disorders of consciousness. It includes three subscales (motor, verbal, and facial responses). Scores range from 0 to 9, with higher scores indicating greater responsiveness to nociceptive stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Estraneo, MD, Principal Investigator — Fondazione Don Gnocchi; Olivia Gosseries, PhD, Professor, Principal Investigator — University of Liege
Locations (2):
- Coma Science Group - University of Liege, Liège, Belgium, Belgium
- Fondazione Don Gnocchi, Sant'Angelo dei Lombardi, Avellino, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD collected throughout the trial (CRS-R, NCS-R, video recordings outcomes, fNIRS data)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the first patient recording data until the last patient.